CLINICAL TRIAL: NCT07401654
Title: Exploratory Study on the Efficacy and Safety of Paclitaxel Monotherapy Versus Paclitaxel-Carboplatin Combination as Neoadjuvant Chemotherapy in Advanced Ovarian Cancer With High PARK2 Expression
Brief Title: The Efficacy and Safety of Paclitaxel Monotherapy Versus Paclitaxel-Carboplatin Combination as Neoadjuvant Chemotherapy in Advanced Ovarian Cancer With High PARK2 Expression
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-929-01
Record Dates: First submitted 2026-01-14; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Neoadjuvant chemotherapy; Paclitaxel; Carboplatin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel (Experimental): Paclitaxel 175mg/m2 intravenous infusion, repeated every 21 days, for 3 to 4 courses
  Interventions: Drug: Paclitaxel
- Paclitaxel + Carboplatin (Active Comparator): Paclitaxel 175mg/m2 intravenous infusion; followed by carboplatin AUC 5~6 intravenous infusion; repeated every 21 days, for 3~4 courses
  Interventions: Drug: Paclitaxel + Carboplatin

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 175mg/m2 administered intravenously, repeated every 21 days, for 3 to 4 cycles
  Arms: Paclitaxel
Drug: Paclitaxel + Carboplatin — Paclitaxel 175mg/m2 intravenous infusion; followed by carboplatin AUC 5~6 intravenous infusion; repeated every 21 days, for 3~4 courses.
  Arms: Paclitaxel + Carboplatin

SUMMARY:
Platinum-based neoadjuvant chemotherapy (NACT) followed by interval debulking surgery is a crucial treatment paradigm for advanced ovarian cancer. It can reduce tumor burden, increase the rate of R0 resection, and decrease surgical complications. The combination of paclitaxel and carboplatin is the standard NACT regimen for ovarian cancer; however, it has limitations: 1) The myelotoxicity of platinum agents may disrupt treatment continuity, and 2) Platinum-based NACT often induces the earlier development of platinum resistance. Therefore, there is a need to explore novel regimens that, while maintaining therapeutic efficacy, can reduce drug exposure and toxicity, delay platinum exposure, and postpone the onset of platinum resistance.

Previous research has revealed that PARK2 can degrade phosphorylated BCL2, thereby enhancing sensitivity to paclitaxel. We established a PARK2-based molecular classification and found that 57% of advanced ovarian cancer cases exhibit high PARK2 expression. Furthermore, ovarian cancers with high PARK2 expression are highly sensitive to paclitaxel. In these patients, a platinum-free paclitaxel regimen demonstrated superior progression-free survival compared to paclitaxel-platinum combination therapy. Based on these findings, we hypothesize that for PARK2-high advanced ovarian cancer, neoadjuvant chemotherapy with single-agent paclitaxel could reduce toxicity and delay premature platinum exposure while achieving efficacy comparable to the standard doublet regimen.

To test this scientific hypothesis, our team plans to conduct an exploratory clinical study. We will enroll patients with advanced, treatment-naive, surgically unresectable, PARK2-high ovarian cancer and randomize them into two cohorts: one receiving neoadjuvant single-agent paclitaxel and the other receiving neoadjuvant paclitaxel plus carboplatin. The study aims to evaluate the efficacy and safety of single-agent paclitaxel NACT in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-75 years.
* Histologically confirmed FIGO Stage III-IV high-grade serous or endometrioid ovarian cancer, primary peritoneal cancer, or fallopian tube cancer via laparotomy, laparoscopy, or core needle biopsy.
* Presence of at least one measurable lesion on CT/MRI, meeting at least one of the following conditions:

  * Failure to achieve R0 cytoreduction (Fagotti score ≥ 8 or upper abdominal CT score ≥ 3).
  * Presence of factors indicating surgical intolerance (meeting ≥1 item): Age ≥75 years; BMI ≥40; Chronic underlying diseases; Malnutrition or hypoalbuminemia; Moderate to large volume ascites; Newly diagnosed venous thromboembolism; ECOG performance status >2.
* High expression of the PARK2 gene in both tumor tissue and blood (Spatial Imaging [SI] score in tumor tissue ≥ 7).
* Expected survival time > 12 weeks.
* ECOG performance status of 0-2.
* Adequate organ function meeting the following criteria:

  * Bone Marrow Function: Absolute neutrophil count (ANC) ≥ 1,500/mm³ (1.5 × 10⁹/L); Platelet count ≥ 100,000/mm³ (100 × 10⁹/L); Hemoglobin ≥ 10 g/dL (100 g/L).
  * Liver Function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); Direct bilirubin ≤ 1 × ULN; AST/ALT ≤ 2.5 × ULN (≤ 5 × ULN if liver metastases are present).
  * Renal Function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula).
* For women of childbearing potential:

  * Negative pregnancy test within 1 week prior to enrollment.
  * Agreement to use effective non-hormonal contraception (e.g., barrier method/intrauterine device) during the study period.
  * Not currently breastfeeding.
* Recovery from prior chemotherapy-related toxicities to ≤ Grade 1 per CTCAE (or baseline level), except for stable sensory neuropathy or alopecia (which may be ≤ Grade 2).
* Willingness to provide tissue and blood samples during the treatment period.
* Ability to understand and voluntarily comply with the study protocol requirements, including:

  * Adherence to the prescribed treatment schedule.
  * Completion of required laboratory tests and imaging assessments per protocol.
  * Participation in the planned follow-up procedures.
* Willingness to complete quality of life questionnaire assessments.

Exclusion Criteria:

* Individuals involved in the planning or conduct of this study.
* Patients concurrently participating in other clinical trials, using other investigational drugs, or receiving neoadjuvant therapies (chemotherapy/radiotherapy/immunotherapy/traditional Chinese medicine therapy).
* Known hypersensitivity or allergy to paclitaxel or carboplatin.
* Patients with dysphagia or gastrointestinal disorders that could affect drug absorption, distribution, metabolism, or excretion (ADME).
* Active symptomatic brain metastases requiring surgery, radiation, and/or corticosteroid therapy, or patients with clinical signs of spinal cord compression.
* Major surgery within 3 weeks prior to study initiation without full recovery.
* Previous or current diagnosis of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or other primary malignancies (except for adequately treated basal cell or squamous cell carcinoma of the skin, ductal carcinoma in situ of the breast, or carcinoma in situ of the cervix).
* Diseases or conditions associated with a high risk of toxicity, including:

  * HIV infection, active hepatitis B or C.
  * Severe cardiovascular diseases (e.g., refractory ventricular arrhythmia, myocardial infarction within the past 3 months).
  * Uncontrolled grand mal seizures, unstable spinal cord compression, or superior vena cava syndrome.
  * Psychiatric illness that would impair the patient's ability to provide informed consent.
  * Uncontrolled hypertension or any other condition deemed by the investigator to be unsuitable for study participation.
  * Prior medical history or existing clinical conditions that may interfere with the interpretation of study results or patient compliance.
  * Transfusion of platelets or red blood cells within 3 days prior to the start of study drug administration.
  * Unresolved clinical toxicities ≥ Grade 2 (except for neuralgia, lymphopenia, and skin depigmentation).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a chemotherapy reaction score of 3 (CRS3) | Perioperative/Periprocedural
Incidence of grade 3-4 neutropenia | During the 2-year follow-up period, from the start of randomization to the patient's withdrawal from the study

SECONDARY OUTCOMES:
Satisfactory tumor reduction rate | Perioperative/Periprocedural
R0 resection rate | Perioperative/Periprocedural
Surgical complexity | Perioperative/Periprocedural
  The measurement that will be used to assess this outcome measure is the Aletti Surgical Complexity Score (SCS), also known as the Surgical Complexity Scoring System for advanced ovarian cancer. This validated scoring system quantifies the complexity of cytoreductive surgery by assigning a weighted point value to specific surgical procedures performed within three anatomical compartments (upper abdomen, mid abdomen, and pelvis). Procedures such as bowel resection, diaphragmatic surgery, splenectomy, and extensive peritonectomy contribute to a total score, which categorizes the surgical effort as low, intermediate, or high complexity.
Progression-free survival (PFS) | During the 2-year follow-up period, the time elapsed from the start of randomization to disease progression or death
Objective response rate (ORR) | During the 2-year follow-up period, from patient randomization to the tumor volume reduction reaching 30%
Incidence of platinum resistance in first recurrence | After the treatment, the disease recurred within 6 months
Overall survival (OS) | During the 2-year follow-up period, the time elapsed from randomization to death
Quality of Life (QoL) | During the 2-year follow-up period, from the beginning of randomization to the end of the study
  Quality of Life, measured by the European Organisation for Research and Treatment of Life Questionnaire-Core 30 (EORTC QLQ-C30), version 3.0 (score range: 0-100; higher scores in global health status/functional scales indicate better quality of life, whereas higher scores in symptom scales indicate worse symptoms) and the ovarian cancer-specific module 28-item (QLQ-OV28) questionnaire. Data will be collected via paper-based questionnaires before treatment initiation and during treatment, and via paper-based questionnaires or telephone interviews during the survival follow-up period. The assessment will be terminated upon patient death, withdrawal of informed consent, or upon disease recurrence or metastasis (regardless of whether the randomly assigned treatment is discontinued).
Incidence of treatment-related adverse events (TRAEs) | During the 2-year follow-up period, from the time of randomization to the time when the patient was discharged from the study